CLINICAL TRIAL: NCT04895553
Title: Incidence of Intracranial Hemorrhage in Glioma Patients With Venous Thromboembolism Converted From LMWH to Apixaban
Status: Terminated | Type: Observational
Why Stopped: lack of funds. Only 1 patient was enrolled
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: ABTCv2-2102; IRB00242129 (Other: Johns Hopkins); J2026 (Other: Johns Hopkins)
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Glioma, Malignant
Keywords: Apixaban; Glioma; ICH; DVT; LMWH
MeSH Terms: conditions — Glioma | interventions — vinyltriethoxysilane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort Apixaban: patients who have switched from low molecular weight heparin (LMWH) to apixaban at the recommended dose of the treating physician.
  FDA approved dose 10 mg twice daily (BID) for 7 days followed by 5 mg PO BID OR physician prescribed dose
  Interventions: Other: Observation of ICH and VTE

INTERVENTIONS:
Other: Observation of ICH and VTE — The treating physician will initiate and prescribe the apixaban, the protocol will only observe and record intracranial pressure (ICP) and VTE incidences.

SUMMARY:
Glioma patients with history of venous thromboembolism (VTE) treated on low molecular weight heparin (LMWH) and who decided with their physician to convert to Apixaban (oral drug) will be enrolled into our study and will collect data regarding recurrent VTE and Intracranial hemorrhage and the incidence of these events.

DETAILED DESCRIPTION:
Primary Objectives To estimate the incidence of intracranial hemorrhage (ICH) in glioma patients with history of venous thromboembolism (VTE) after the conversion from low molecular weight heparin (LMWH) injections to oral Apixaban.

Secondary Objective To estimate the incidence of recurrent VTE in glioma patients with history of venous thromboembolism after the conversion from low molecular weight heparin (LMWH) injections to oral Apixaban.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older;
* Patients must have had a pathologically confirmed supra-tentorial primary brain tumor
* Patients must have history of deep venous thrombosis (DVT) and/or pulmonary embolism (PE)
* Patients must have been treated with low molecule weight heparin for ≥ 5 days
* Patients must be able to provide written informed consent
* Patients must have non contrast CT that is negative for intra-cranial bleed at least 5 days post initiation of LMWH and prior to initiation (within 7 days) of Apixaban
* Must be decision by patient and his physician to convert to Apixaban

Exclusion Criteria:

* Patients with a plan less than 6 months of anticoagulation for most recent DVT or PE
* Patients with allergic reaction to Apixaban
* Patients with active bleeding or high risk for bleeding contraindicating treatment with LMWH
* Patients with planned surgery in the next 2 weeks
* Patients previously treated with Apixaban
* Patients requiring Acetylsalicylic Acid (ASA) greater than165 mg/day at enrollment
* Patients requiring dual anti-platelet therapy (ASA plus clopidogrel or ASA plus ticlopidine) at enrollment.
* Subjects with transition for dual anti-platelet therapy or monotherapy prior to enrollment will be eligible for the study
* Patients who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness
* Any condition, which in the opinion of the investigator, would put the subject at an unacceptable risk from participating in the study
* Any other medical, social, logistical, or psychological reason, which in the opinion of the investigator, would preclude compliance with, or successful completion of, the study protocol
* Known active and clinically significant liver disease (e.g., hepatorenal syndrome)
* Known bacterial endocarditis
* Know uncontrolled hypertension: systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg; (subjects who have a transient, higher blood pressure elevation associated with acute PE [upper limit: systolic blood pressure 200 mm Hg or diastolic blood pressure 100 mm Hg] may enter the study;) elevated blood pressure that is persistent 1 - 2 days after the index DVT or PE should be treated according to local guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients greater than or equal to 18 years of age who have had a pathologically confirmed supra-tentorial primary brain tumor and a history of deep venous thrombosis (DVT) and/or pulmonary embolism (PE).
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Intracranial Hemorrhage (ICH) event incidence rate | 1 year
  Observe subject to determine the incidence of ICH during standard of care (SOC) observations.

SECONDARY OUTCOMES:
Deep venous thromboembolism (VTE) event incidence rate | 1 year
  Observe subject to determine the incidence of VTE during SOC observations.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Grossman, MD, Study Chair — Johns Hopkins University
Locations (2):
- United States (2):
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Johns Hopkins, Baltimore, Maryland